CLINICAL TRIAL: NCT06153745
Title: Aspheric Monofocal Intraocular Lens With Higher Order Aspheric Optic in Pediatric Patients: Early Outcomes
Brief Title: Aspheric Monofocal Intraocular Lens in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Luca Buzzonetti (Other)
Responsible Party: Sponsor-Investigator, Luca Buzzonetti, Head of Ophthalmology Unit, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Other Study IDs: BG123
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Cataract in Child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tecnis Eyhance ICB00 intraocular lens (Johnson&Johnson Vision, Santa Ana, California USA) — pediatric cataract surgery

SUMMARY:
To evaluate the performance a new aspheric monofocal intraocular lens (IOL) with higher order aspheric optic for far, intermediate, and near vision, in pediatric patients after monolateral cataract surgery.

DETAILED DESCRIPTION:
thirteen patients (mean age 7.6±3.8 years) who underwent cataract surgery and simultaneous implantation of the Tecnis Eyhance ICB00 IOL were evaluated. Visual acuity was assessed three months after surgery for distance (CDVA), intermediate (CIVA) and near visual acuity (CNVA).

ELIGIBILITY:
Inclusion Criteria:

* monolateral cataract

Exclusion Criteria:

* other ocular diseases
* systemic diseases

Ages: 6 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Corrected Distance Visual Acuity | 3 months postoperatively
  Decimal
Corrected Intermediate Visual Acuity | 3 months postoperatively
  Decimal
Corrected Near Visual Acuity | 3 months postoperatively
  Decimal

CONTACTS AND LOCATIONS:
Overall Officials: Luca Buzzonetti, Principal Investigator — Bambino Gesù Children's Hospital, Rome, Italy
Locations (1):
- Luca Buzzonetti, Roma, Italy